CLINICAL TRIAL: NCT01375205
Title: A Randomized Pilot Trial Comparing Cetaphil® Restoraderm® System and Standard Skin Care in Infants at Risk for Atopic Dermatitis
Brief Title: Comparing Cetaphil Restoraderm System Versus Standard Skin Care in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Eric Simpson, M.D., M.C.R., Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Galderma Cetaphil Restoraderm
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; skin care
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Standard of Care; Ad26COVS1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Active Comparator): Subjects will apply Johnson&Johnson moisturizer to their infant's skin as often as they wish. They will also use the Johnson&Johnson cleanser.
  Interventions: Other: Standard of Care
- Cetaphil Restoraderm (Experimental): Subjects will apply Cetaphil Restoraderm moisturizer once daily to infant's skin. They will bathe their infant with Cetaphil Restoraderm cleanser.
  Interventions: Other: Cetaphil Restoraderm

INTERVENTIONS:
Other: Cetaphil Restoraderm — Subjects will apply Cetaphil Restoraderm moisturizer once daily to infant's skin. They will bathe their infant with Cetaphil Restoraderm cleanser.
  Arms: Cetaphil Restoraderm
Other: Standard of Care — Subjects will apply Johnson&Johnson moisturizer to their infant's skin as often as they wish. They will also use the Johnson&Johnson cleanser.
  Other Names: Johnson&Johnson
  Arms: Standard of Care

SUMMARY:
The goal of this study is to determine what effect Cetaphil® Restoraderm® system has on babies' skin versus Johnson & Johnson baby lotion and skin cleanser.

DETAILED DESCRIPTION:
Subjects will randomly be divided into a group using Cetaphil® Restoraderm® system or a group using Johnson & Johnson baby lotion and skin cleanser . At 3, 6, and 12 months non-invasive measurements of barrier function will be used to test the babies' skin. The procedures are as follows:

* Transepidermal loss (TEWL - measures the water loss from the skin)
* Skin electrical capacitance (measures how much water stays in the top layer of skin)
* Skin pH (measures level of pH)
* Skin microbiome analysis (skin swabs to check genetic code of skin bacteria)
* Lipidomic and natural moisturizing factor analysis (measures lipids (oils) in the top layer of skin)

Both groups will be reminded to follow the instructions about general good skin care of infants. Subjects will be asked if they agree to provide a saliva sample. If yes, a saliva sample will be collected from the inside of the infant's cheek at the 6 month visit and will be shipped to the laboratory of Dr. Irwin McLean at the University of Dundee, where it will be tested for gene defects in the skin barrier that might trigger the development of eczema. Defects in the gene called filaggrin have been shown to increase the risk of developing eczema. The samples will be identified by a code to protect your infant's identity. The saliva samples will be stored only for this study, and then the sample will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Infants up to three weeks of age born to mothers aged 18-45 years will be recruited for this study.
* Infants must have a family history of asthma, eczema, or hayfever in at least one first-degree relative and be in otherwise good overall health.

Exclusion Criteria:

* Preterm birth defined as birth prior to 37 weeks gestation
* Major congenital anomaly
* Hydrops fetalis
* Significant dermatitis at birth not including seborrheic dermatitis on the scalp ("cradle cap")
* Any immunodeficiency disorder
* Any severe genetic skin disorder
* Any other serious condition that would make the use of emollients inadvisable
* Any other major medical problems that the investigator deems may increase the risk of adverse events with the intervention or in whom assessing the outcomes may be masked by the underlying problem or practically very difficult to assess

Ages: 1 Day to 3 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Simpson, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University Center for Health & Healing, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetaphil Restoraderm | Standard of Care
Started | 54 | 46
Completed | 33 | 33
Not Completed | 21 | 13
Not completed — Lost to Follow-up | 15 | 12
Not completed — Withdrawal by Subject | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetaphil Restoraderm | Standard of Care | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 46 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 30 | 21 | 51
Region of Enrollment [Number; unit: participants]
  United States | 54 | 46 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cumulative Atopic Dermatitis Diagnosed by Investigator at 12 Months
Description: Percentage of cumulative Atopic Dermatitis diagnosed by a blinded investigator at 12 months
Time Frame: 12 months
Population: Around 28% of subjects enrolled were lost to follow-up by 12 months
Measure: Number; unit: Percentage of participants
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 38 | 32
Percentage of participants | 13.2 | 25

2. Secondary Outcome: Percentage of High Emollient Use
Description: Patient-reported adherence to the emollient regimen in the intervention group and the treatment group. High emollient use was defined as applying the intervention or control emollient five or more days per week.
Time Frame: 2, 6, 12, 18, and 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 54 | 46
percentage of participants
  Percentage of high emollient use at 2 months | 87 | 45.2
  Percentage of high emollient use at 6 months | 72.4 | 45.8
  Percentage of high emollient use at 12 months | 66.7 | 45.5
  Percentage of high emollient use at 18 months | 52.2 | 53.3
  Percentage of high emollient use at 24 months | 40.0 | 33.3

3. Secondary Outcome: Age at Onset of Eczema
Description: Age of subject at onset of eczema
Time Frame: Baseline through Month 24 Follow-up
Measure: Median (Full Range); unit: months
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 54 | 46
months | 4 [0 to 24] | 6 [0 to 24]

4. Secondary Outcome: Filaggrin Mutation Status
Description: Filaggrin mutation status result
Time Frame: 6 month visit
Population: Number of participants analyzed captures only those participants that completed 6 month filaggrin testing. Not all participants noted in the overall participant flow were able to complete filaggrin testing either due to study status (i.e., lost to follow up, withdrawn) or missed visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 25 | 31
Participants
  Positive for Filaggrin Mutation | 3 | 2
  Negative for Filaggrin Mutation | 22 | 29

5. Secondary Outcome: Transepidermal Water Loss (TEWL)
Description: Transepidermal water loss (TEWL) to measure skin barrier function
Time Frame: 2 month, 6 month, and 12 month visits
Population: Number of participants analyzed captures only those participants that completed TEWL testing at all time points. Not all participants noted in the overall participant flow were able to complete TEWL testing either due to study status (i.e., lost to follow up, withdrawn) or missed visits.
Measure: Mean (Standard Deviation); unit: (g/[m2hr])
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 32 | 24
(g/[m2hr])
  Average TEWL (g/[m2hr]) at 2 months | 16.3 (7.1) | 18.3 (8.6)
  Average TEWL (g/[m2hr]) at 6 months | 15.9 (5.6) | 16.1 (6.2)
  Average TEWL (g/[m2hr]) at 12 months | 13.9 (2.3) | 16.7 (5.6)

6. Secondary Outcome: Skin Hydration (Skin Electrical Capacitance)
Description: Determination of stratum corneum hydration from the dorsal forearm
Time Frame: 2 month, 6 month, and 12 month visits
Population: Number of participants analyzed captures only those participants that completed skin hydration testing at all time points. Not all participants noted in the overall participant flow were able to complete skin hydration testing either due to study status (i.e., lost to follow up, withdrawn) or missed visits.
Measure: Mean (Standard Deviation); unit: farads
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 32 | 24
farads
  Average capacitance at 2 months | 55.2 (14.0) | 53.9 (8.2)
  Average capacitance at 6 months | 51.8 (9.8) | 52.1 (6.1)
  Average capacitance at 12 months | 49.4 (12.7) | 53.7 (14.0)

7. Secondary Outcome: Skin pH
Description: Skin pH, as measured using a pH probe
Time Frame: 2 month, 6 month, and 12 month visits
Population: Number of participants analyzed captures only those participants that completed Skin pH testing at all time points. Not all participants noted in the overall participant flow were able to complete Skin pH testing either due to study status (i.e., lost to follow up, withdrawn) or missed visits.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 32 | 24
pH
  Average pH at 2 months | 5.5 (0.4) | 5.2 (0.4)
  Average pH at 6 months | 5.3 (0.6) | 5.4 (0.5)
  Average pH at 12 months | 5.4 (0.7) | 5.4 (0.5)

8. Post Hoc Outcome: Percentage of Participants With Cumulative Atopic Dermatitis Diagnosed by Investigator at 24 Months
Description: Percentage of cumulative Atopic Dermatitis diagnosed by any MD at 24 Months
Time Frame: 24 Months
Population: Number of participants analyzed captures only those participants still on study at 24 months.
Measure: Number; unit: percentage of participants
Arm/Group | Cetaphil Restoraderm | Standard of Care
Number analyzed (Participants) | 31 | 29
percentage of participants | 19.4 | 31.0

ADVERSE EVENTS:
Time Frame: From the time informed consent is signed through the 24 month study follow-up telephone call.
Arm/Group | Cetaphil Restoraderm | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/54 | 0/46
Other Adverse Events (participants affected / at risk) | 30/54 | 21/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetaphil Restoraderm (N=54) | Standard of Care (N=46)
Idiopathic Intracranial Hypertension (Nervous system disorders) | 1 (1) | 0 (0)
RSV and Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetaphil Restoraderm (N=54) | Standard of Care (N=46)
Baby Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Viral exanthems (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Heat rash/miliaria (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Candidiasis (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8)
Diaper dermatitis (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)
Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (8)
Bacterial Skin Infection (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Unspecified Transient Rashes (Skin and subcutaneous tissue disorders) | 9 (9) | 3 (3)
Rash to Vaccination/Drug Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Irritant Contact Dermatitis (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Urticarial Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No